CLINICAL TRIAL: NCT01604772
Title: A Phase II Study of MK-2206 in Patients With Progressive, Recurrent/Metastatic Adenoid Cystic Carcinoma
Brief Title: Akt Inhibitor MK2206 in Treating Patients With Progressive, Recurrent, or Metastatic Adenoid Cyst Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01966; NCI-2012-01966 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000733948; CALGB-A091104; A091104 (Other: Alliance for Clinical Trials in Oncology); A091104 (Other: CTEP); N01CM62206 (NIH); R01CA166978 (NIH); U10CA180821 (NIH); U10CA031946 (NIH)
Record Dates: First submitted 2012-05-22; First posted 2012-05-24 (Estimated); Results first posted 2015-06-26 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Recurrent Oral Cavity Adenoid Cystic Carcinoma; Recurrent Salivary Gland Carcinoma; Salivary Gland Adenoid Cystic Carcinoma; Stage IVA Major Salivary Gland Cancer AJCC v7; Stage IVA Oral Cavity Adenoid Cystic Carcinoma AJCC v6 and v7; Stage IVB Major Salivary Gland Cancer AJCC v7; Stage IVB Oral Cavity Adenoid Cystic Carcinoma AJCC v6 and v7; Stage IVC Major Salivary Gland Cancer AJCC v7; Stage IVC Oral Cavity Adenoid Cystic Carcinoma AJCC v6 and v7
MeSH Terms: conditions — Salivary Gland Neoplasms | interventions — MK 2206

ARMS (1):
- Treatment (Akt inhibitor MK2206) (Experimental): Patients receive Akt inhibitor MK2206 PO once weekly for 4 weeks. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Akt Inhibitor MK2206; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Akt Inhibitor MK2206 — Given PO
  Other Names: MK2206
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well Akt inhibitor MK2206 works in treating patients with progressive, recurrent, or metastatic adenoid cyst carcinoma (cancer). Akt inhibitor MK2206 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the confirmed response rate of patients with progressive, recurrent/metastatic adenoid cyst carcinoma (ACC) treated with v-akt murine thymoma viral oncogene homolog 1 (Akt) inhibitor MK2206 (MK-2206).

SECONDARY OBJECTIVES:

I. To evaluate the progression-free survival (PFS), overall survival (OS), and safety/tolerability for MK-2206 in these patients.

TERTIARY OBJECTIVES:

I. To explore potential genetic/cytogenetic/histopathologic predictors of clinical outcome (i.e., response, PFS, OS) to MK-2206.

II. To explore the hypothesis that MK-2206-mediated Akt inhibition and downregulation of v-myb avian myeloblastosis viral oncogene homolog (c-myb) protein levels in ACC tumors correlates to clinical outcome (i.e., response, PFS, OS).

OUTLINE:

Patients receive Akt inhibitor MK2206 orally (PO) once weekly for 4 weeks. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of treatment, patients are followed up every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically confirmed adenoid cystic carcinoma; confirmation will be performed locally at each participating institution; cancers arising from non-salivary gland primary sites are allowed
* Patients must have measurable disease, as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 2.0 cm with conventional techniques or as >= 1.0 cm with spiral computed tomography (CT) scan; to be considered pathologically enlarged and measurable, a lymph node must be > 1.5 cm in short axis when assessed by CT scan (CT scan slice-thickness recommended to be no greater than 5 mm)
* Patients must have locally advanced and/or recurrent and/or metastatic disease not amenable to potentially curative surgery or radiotherapy
* Patients must have increasing disease, defined as the presence of new or progressive lesion(s) on CT/magnetic resonance imaging (MRI) within 6 months prior to study enrollment and/or new/worsening disease-related symptoms; NOTE: this increase in disease is to be determined in the oncologist's best judgment and does not have to meet Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* Chemotherapy and radiation therapy must be completed at least 4 weeks prior to registration; if the last regimen included Carmustine (BCNU) or mitomycin C, it must be completed at least 6 weeks prior to registration; NOTE: any number of prior chemotherapy regimens is allowed, including no prior treatment
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (equivalent to Karnofsky >= 50%)
* Leukocytes >= 3,000/mm^3
* Absolute neutrophil count >= 1,000/mm^3
* Platelets >= 75,000/mm^3
* Total bilirubin =< institutional upper limit of normal (ULN)
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) or serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 2.5 institutional upper limit of normal
* Creatinine =< ULN OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above ULN
* Patients must be able to swallow whole tablets; NOTE: nasogastric or gastric (G) tube administration is not allowed; tablets must not be crushed or chewed
* Patients must have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have received prior treatment with phosphatidylinositol-4,5-bisphosphate 3-kinase, catalytic subunit alpha (PI3K), v-akt murine thymoma viral oncogene homolog 1 (Akt), or mechanistic target of rapamycin (serine/threonine kinase) (mTOR) inhibitors for recurrent/metastatic ACC
* Patients who are receiving any other investigational agents
* Patients with known brain metastases
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MK-2206 or other agents used in the study
* Patients receiving any medications or substances that are major inhibitors or inducers of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP450 3A4)
* Diabetic patients with glycated hemoglobin (HbA1c) levels of greater than 8%; NOTE: preclinical studies demonstrated the potential of MK-2206 for induction of hyperglycemia in all preclinical species tested; patients with diabetes or at risk for hyperglycemia should not be excluded from trials with MK-2206, but the hyperglycemia should be well controlled before the patient enters the trial
* Cardiovascular baseline Fridericia corrected QT (QTcF) > 450 msec (male) or QTcF > 470 msec (female) will exclude patients from entry on study; NOTE: medications that may cause QTc interval prolongation should be avoided by patients entering on trial
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirements
* Pregnant women; NOTE: women of child-bearing potential must have a negative serum or urine pregnancy test within 7 days prior to registration

  * Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
  * Breastfeeding should be discontinued if the mother is treated with MK-2206
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy
* Other active malignancy, other than indolent malignancies which the investigator determines are unlikely to interfere with treatment and safety analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-07-23 (Actual); Primary Completion 2013-10-24 (Actual); Study Completion 2014-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Ho, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (51):
- United States (51):
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Reid Health, Richmond, Indiana
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Union Hospital of Cecil County, Elkton, Maryland
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Carolinas HealthCare System NorthEast, Concord, North Carolina
  - Carolinas HealthCare System Union, Monroe, North Carolina
  - Carolinas HealthCare System Cleveland, Shelby, North Carolina
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Ho AL, Foster NR, Deraje Vasudeva S, Katabi N, Antonescu CR, Frenette GP, Pfister DG, Erlichman C, Schwartz GK. A phase 2 study of MK-2206 in patients with incurable adenoid cystic carcinoma (Alliance A091104). Cancer. 2024 Mar 1;130(5):702-712. doi: 10.1002/cncr.35103. Epub 2023 Nov 10. PMID 37947157

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Akt Inhibitor MK2206): Patients receive Akt inhibitor MK2206 PO once weekly for 4 weeks. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Akt Inhibitor MK2206: 150 mg given PO
Period: Overall Study
Arm/Group | Treatment (Akt Inhibitor MK2206)
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 16
Age, Continuous [Median (Full Range); unit: years] | 63.5 [31 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Response Rate (Complete Response + Partial Response) According to RECIST Version 1.1
Description: Confirmed response rate will be reported as the number of participants achieving either a complete response or partial response (using RECIST v1.1) divided by the number of evaluable participants. In order for a participant to be a confirmed objective responder, they must achieve a PR or CR on consecutive evaluations, at least 4 weeks apart.
  Complete Response (CR): Disappearance of all target lesions and normalization of tumor biomarkers.
  Partial Response (PR): At least a 30% decrease in the sum of the LD of target lesions taking as reference the baseline sum LD.
Time Frame: Up to 32 weeks
Population: Two patients were deemed ineligible for this endpoint due to eligibility criteria not being met. Therefore, this endpoint is reported using 14 eligible patients.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 14
percentage of patients | 0 [0 to 23.2]

2. Secondary Outcome: Median Progression Free Survival
Description: Progression Free Survival is defined as the time from registration to the earliest date of documentation of disease progression or death. The distribution of time to progression will be estimated using the method of Kaplan-Meier.
Time Frame: Time of study entry to progression or death, up to 3 years after registration
Population: Two patients were deemed ineligible and were not included in this endpoint.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 14
months | 9.7 [3.8 to 11.8]

3. Secondary Outcome: Overall Survival
Description: Overall Survival is defined as the time from registration to death. The distribution of survival will be estimated using the method of Kaplan-MeierEstimated using Kaplan-Meier methodology.
Time Frame: Time of study entry to death due to any cause, assessed up to 3 years from registration
Population: Two patients were not eligible for this endpoint.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 14
months | 18 [11.8 to 29.9]

4. Secondary Outcome: Incidence of Toxicities of Akt Inhibitor MK-2206
Description: Safety will be assessed in terms of the number of participants reporting grade 3 or higher adverse events as evaluated by Common Terminology Criteria for Adverse Events v4.0 (CTCAE).
Time Frame: Time to first treatment to up to 30 days after completion of treatment
Population: All patients that started protocol treatment were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 16
Participants
  Grade 3 Adverse Event | 10
  Grade 4 Adverse Event | 2

ADVERSE EVENTS:
Arm/Group | Treatment (Akt Inhibitor MK2206)
Serious Adverse Events (participants affected / at risk) | 2/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Akt Inhibitor MK2206) (N=16)
Esophageal hemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Akt Inhibitor MK2206) (N=16)
Anemia (Blood and lymphatic system disorders) | 3 (12)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 6 (14)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (3)
Eye disorders - Other, specify (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Cheilitis (Gastrointestinal disorders) | 1 (10)
Constipation (Gastrointestinal disorders) | 2 (10)
Diarrhea (Gastrointestinal disorders) | 4 (10)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 3 (4)
Nausea (Gastrointestinal disorders) | 4 (6)
Oral pain (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 13 (38)
Pain (General disorders) | 2 (3)
Bronchial infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (3)
Fall (Injury, poisoning and procedural complications) | 1 (3)
Alanine aminotransferase increased (Investigations) | 2 (6)
Alkaline phosphatase increased (Investigations) | 2 (11)
Aspartate aminotransferase increased (Investigations) | 1 (3)
Creatinine increased (Investigations) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 2 (2)
Investigations - Other, specify (Investigations) | 1 (4)
Lymphocyte count decreased (Investigations) | 7 (12)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 7 (29)
Weight loss (Investigations) | 5 (22)
White blood cell decreased (Investigations) | 1 (10)
Anorexia (Metabolism and nutrition disorders) | 6 (15)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 14 (51)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (5)
Hypernatremia (Metabolism and nutrition disorders) | 2 (3)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (6)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3)
Dysgeusia (Nervous system disorders) | 2 (8)
Headache (Nervous system disorders) | 2 (10)
Memory impairment (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (10)
Anxiety (Psychiatric disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (6)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (10)
Purpura (Skin and subcutaneous tissue disorders) | 1 (6)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 13 (58)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 (13)
Hypertension (Vascular disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less